CLINICAL TRIAL: NCT03772275
Title: Clinical and Economical Study Evaluating the Utility of Some Novel Biomarkers of Patients With Chronic Heart Failure
Brief Title: Utility of Some Novel Biomarkers of Patients With Chronic Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Heart failure
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New york Heart Association Class II-IV (Active Comparator): New york Heart Association Class II-IV heart failure
  Interventions: Diagnostic Test: New york Heart Association Class II-IV
- New york Heart Association Class I (Active Comparator): New york Heart Association Class I with no heart failure
  Interventions: Diagnostic Test: New york Heart Association Class I

INTERVENTIONS:
Diagnostic Test: New york Heart Association Class II-IV — New york Heart Association Class II-IV " study of markers"
  Other Names: Severe heart failure
  Arms: New york Heart Association Class II-IV
Diagnostic Test: New york Heart Association Class I — New york Heart Association Class I
  Other Names: No heart failure
  Arms: New york Heart Association Class I

SUMMARY:
Clinical and Economic study of some new biomarkers in chronic heart failure.

DETAILED DESCRIPTION:
The study aimed at evaluation of the clinical and economic value of some new biomarkers in chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* NYHA-Class II-IV

Exclusion Criteria:

* Liver or renal dysfunction. --DM

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with elevated markers (IL17) | 6 months
  Number of participants with elevated markers (IL17)

CONTACTS AND LOCATIONS:
Overall Officials: Osama M Ibrahim, Prof, Principal Investigator — Prof of Clinical Pharmacy; Medhat M Eshmawy, Prof, Study Director — Cardiology Department- Tanta University; Nermin W Ishaq, Msc, Study Chair — Clinical pharmacy Department- Tanta University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided